CLINICAL TRIAL: NCT05293821
Title: A Multicenter Clinical Performance Study to Compare the Results Obtained From the TriQuik Invitro Diagnostic Device With Historical Medical Records From the Same Subject
Brief Title: Multicenter Performance Study of TriQuik Invitro Diagnostic Device
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Genlantis Diagnostics (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Robert Zeiler, Chief Scientific Officer, Genlantis Diagnostics
Other Study IDs: GENL-TQ 002
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-03

CONDITIONS: To Demonstrate Clinical Performance of the TriQuik Invitro Diagnostic Device
Keywords: TriQuik IVD, HIV, hepatitis B, hepatitis C
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Positive test subjects: documented medical history of HIV, HBV or HCV. A combination of 2 or 3 conditions is acceptable.
  Interventions: Diagnostic Test: TriQuik IVD
- Control: no documented medical history of HIV, HBV or HCV and are considered normal.
  Interventions: Diagnostic Test: TriQuik IVD

INTERVENTIONS:
Diagnostic Test: TriQuik IVD — TriQuik Invitro Diagnostic Device Cassettes. TriQuik Invitro Diagnostic Device Cassettes.

SUMMARY:
This prospective and historical clinical study is designed to test the performance of the Genlantis TriQuik test kit (Cassette). The primary goal is to establish the sensitivity and specificity (i.e. how accurate the test is) when compared to the same patient's medical history.

Previous tests were performed on serum and whole blood specimens. A total of 607 serum specimens1 were collected for evaluation and comparison of the performance of the TriQuik Hepatitis B Surface Antigen (HBsAg) Test with a licensed commercial HBsAg EIA. 84 of 85 positive serum samples testing by the licensed commercial HBsAg EIA were reactive with TriQuik HBsAg Test and 520 of 522 negative samples testing by the licensed commercial HBsAg EIA were tested negative with TriQuik HBsAg Test.

DETAILED DESCRIPTION:
Study Objective To demonstrate clinical performance of the TriQuik Invitro Diagnostic device.

Measurement Methodology Whole blood samples are collected by fingerstick. Samples should be tested immediately.

Using the supplied sample dropper, transfer specimen blood drop into the sample well. Wait 20-30 seconds. Add two drops of the supplied assay buffer (~90µL) to the same sample well Read result in 20 mins.

Primary end points will determine how accurate these tests are (p<=0.02) by analyzing for:

Diagnostic Sensitivity; TP / (TP + FN) The ability of the test to correctly identify those patients with the disease Diagnostic Specificity; TN / (TN + FP) The ability of the test to correctly identify those patients who are truly free of the specific disease Positive Predictive Value: TP / (TP+ FP) The probability that subjects with a positive test truly have the disease. Negative Predictive Value: TN / (FN + TN) The probability that subjects with a negative test truly don't have the disease.

An estimated 200 patients are to be enrolled as follows:

150 with a documented medical history of HIV, HBV or HCV. A combination of 2 or 3 conditions is acceptable.

HbsAg patients need to have a HbsAg on file < 2 years. HIV and HCV patients only need one antibody test in their medical chart.

50 with no documented medical history of HIV, HBV or HCV and are considered normal.

Male or female subjects, ages ≥18 years.

ELIGIBILITY:
Inclusion Criteria:

* a documented medical history of HIV, HBV or HCV. A combination of 2 or 3 conditions is acceptable.

  * HbsAg patients need to have a HbsAg on file < 2 years.
  * HIV and HCV patients only need one antibody test in their medical chart.
* no documented medical history of HIV, HBV or HCV and are considered normal.
* Male or female subjects, ages ≥18 years.
* Signed informed consent provided by an authorized subject representative (based on local Institutional Review Board (IRB)/ethics panel requirements).

Exclusion Criteria:

Any other condition or prior therapy, which, in the opinion of the investigator, would make the subject unsuitable for this study.

Participation in any phase of another clinical research study involving the evaluation of another investigational drug or device within 30 days before randomization.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study patients are seen, recruited and consented from local clinics and physician offices.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Standard performance criteria | <1 day
  Diagnostic Sensitivity, Diagnostic Specificity, Positive Predictive Value, Negative Predictive Value

IPD SHARING:
Plan to Share IPD: Yes
There will be a need to communicate the results of this clinical performance study to clinicians and/or public health institutions and regulatory bodies after the study. This is the case since these test results have an immediate health impact to the patient, patient's relatives and the public.
  The decision and the mechanism to report results to clinicians and public health institutions will be discussed with the local ethics committee prior to beginning the clinical performance study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Two months following completion of analysis

REFERENCES:
- See also: Related Info — http://www.genlantisdx.com